CLINICAL TRIAL: NCT04540640
Title: Feasibility of Subnormothermic Oxygenated Machine Perfusion for Protection of Renal Allografts: A Single Centre Pilot Study
Brief Title: Oxygenated Machine Preservation in Kidney Transplantation
Acronym: SNOPO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Patrick Luke, Surgical Director of Multi-Organ Transplant, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 116275
Record Dates: First submitted 2020-08-25; First posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Kidney Transplantation
Keywords: Perfusion

STUDY DESIGN:
Intervention Model Description: A pilot study assessing the feasibility of procedures and preliminary safety of study device and perfusion solution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Subnormothermic Perfusion (Experimental): Kidneys retrieved for transplantation will undergo subnormothermic oxygenated perfusion using the study device and perfusion solution for at least 1 hour prior to transplantation into the recipient.
  Interventions: Device: Kidney perfusion pump

INTERVENTIONS:
Device: Kidney perfusion pump — The pulsatile perfusion device will circulate room temperature oxygenated perfusion solution through the donor kidney ex vivo.

SUMMARY:
Kidney transplantation remains the best treatment option for patients with end-stage kidney failure, however, the need for transplantable organs far exceeds the number of acceptable grafts available from deceased donors. In an effort to increase access to transplantation, organs from higher risk donors are being used more frequently. Patients who receive these high risk kidneys are more likely to experience poor outcomes post-transplantation, such as delayed graft function and shorter graft survival than those who receive standard criteria donor kidneys. One way to improve outcomes in these high risk kidneys is to limit the amount of damage donor organs sustain during the transplant process. The current standard of care is storage of the donor organ on ice until the time of transplant, during which the kidney incurs injury from cold and lack of oxygen. Recent research suggests that oxygenated machine perfusion of the organ at room temperature as a storage method can help protect kidneys and improve post-transplant outcomes. This study aims to assess the feasibility and safety of room temperature oxygenated machine perfusion of donor kidneys prior to transplantation. Kidney function will be evaluated with standard clinical parameters and participants will be followed for one-year post-transplantation for their outcomes. Feasibility will be evaluated in terms of trial process such as recruitment rate and ease of implementation of the study intervention. Preliminary safety will be assessed by incidence of graft discard and technical limitations.

DETAILED DESCRIPTION:
Kidney transplantation remains the treatment of choice for patients suffering from end-stage renal disease. To combat the ever-increasing waiting list, higher risk organs, including those from donation after circulatory death (DCD) donors, and older donors are being transplanted more frequently. However, organs from these donors are more susceptible to damage during the transplant procedure known as ischemia-reperfusion injury (IRI) and show worse outcomes post-transplant such as increased rates of primary non-function, delayed graft function and early graft loss. Therefore, strategies to mitigate IRI are of great interest to improve transplant outcomes. One method of interest is modification of organ storage techniques during the transplant process.

The current standard of care for organ preservation is static cold storage or hypoxic hypothermic pulsatile perfusion of the donor organ. Our pre-clinical studies in a porcine DCD transplant model indicate that perfusion at room temperature is capable of significantly reducing kidney inflammation and damage during the transplant process compared to cold storage and normothermic perfusion. While other trials have looked at hypothermic and normothermic perfusion, to the best of our knowledge there has not been a trial to evaluate subnormothermic perfusion of kidneys.

The study intervention will consist of ex vivo perfusion of donor kidneys using a clinical pulsatile pump modified with an oxygen delivery unit developed by our laboratory. Once organs arrive at the transplant centre they will be attached to the pump by the transplant surgery team and/or perfusionist. Prior to placement on pump, a baseline tissue sample of the kidney will be taken via needle core biopsy. Kidneys will be perfused with a preservation solution composed of a bloodless oxygen carrier. Organs will be perfused for 1-10 hours depending on the clinical timeline of the transplant. The kidney will be transplanted into the recipient as per clinical standard. After reperfusion of the kidney in the recipient, another study tissue sample will be collected via needle core biopsy. Pre-implantation and post-perfusion baseline biopsies are performed as clinical standards, but a small sample of the biopsy specimen will be stored for analysis in our laboratory. Study participants (n=15) will be followed for 1 year post-transplant and their graft function will be assessed using standard clinical parameters.

The goal of this study is to determine the feasibility and preliminary safety of subnormothermic perfusion. Feasibility will be assessed by ease of implementation of study procedures and recruitment rate. Safety will be determined from rate of graft discard attributed to study intervention, graft function and technical limitations of the study intervention.

ELIGIBILITY:
Inclusion Criteria (Participant):

* Adult male or females, 18 years or older
* Active on the kidney transplant waiting list

Exclusion Criteria (Participant):

* Patients receiving a multi-organ transplant (e.g. double kidney, kidney-pancreas)
* Patients who are unable/refuse to provide informed consent

Inclusion Criteria (Organ):

* Single kidney from donation after circulatory death (DCD) or donation after brain death (DBD) donor.

Exclusion Criteria (Organ):

* Kidneys from living donors
* Kidneys that would be declined for transplantation under current clinical practice
* Vascular issues precluding placement on a pump

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Eligible versus actual kidney perfusions performed to assess study feasibility | 1 year from start of study
  Ratio of kidneys grafts that are planned to receive the study intervention compared to the actual number of grafts perfused by study device.
Rate of kidney discard or graft failure attributed to the study intervention | From first study intervention to 1 year after last intervention
  Complications related to ex vivo perfusion that result in graft discard prior to transplantation or graft failure post-transplantation will be recorded.

SECONDARY OUTCOMES:
Rate of delayed graft function in study participants | 1 year post-transplantation
  The need for post-transplant dialysis in study participants will be recorded
Degree of ischemia-reperfusion injury by kidney biopsy | 3 months after enrolment of last participant
  Pre and post-implantation kidney biopsies will be graded as per standard histological criteria to assess for ischemia-reperfusion injury
Post-transplant serum creatinine levels to assess graft function | From first study intervention to 1 year after transplantation of final participant
  Serum creatinine levels will be interpreted as per clinical standard, with higher levels indicating poorer graft function
Rate of primary non-function of kidney grafts in study participants | 1 year post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Luke, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No